CLINICAL TRIAL: NCT07264868
Title: Home Neuromodulation for Neurogenic Bladder Management in Spinal Cord Injury: A Hybrid Implementation-Efficacy Trial
Brief Title: Home Neuromodulation for Neurogenic Bladder Management in Spinal Cord Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Argyrios Stampas, MD, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-25-0582; CDMRP-SC240085 (Registry Identifier: CDMRP-eBRAP Log Number)
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Spinal Cord Injury (SCI); Neurogenic Bladder (NB)
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Bilateral iTNS (Experimental): participants will receive one active tibial nerve stimulation (TNS) device and both legs will receive active stimulation
  Interventions: Device: iTNS
- Unilateral iTNS (Active Comparator): participants will receive one active and one sham tibial nerve stimulation (TNS) device. The treatment will only be delivered to the leg with the active device.
  Interventions: Device: iTNS; Device: Sham iTNS
- Sham iTNS (Sham Comparator): participants will receive one one sham tibial nerve stimulation (TNS) device for bilateral use.
  Interventions: Device: Sham iTNS

INTERVENTIONS:
Device: iTNS — The stimulation current will be gradually increased until bilateral toe flexion is achieved, then reduced to just below the motor contraction threshold. A 20 Hz frequency and 200 µs pulse width will be applied continuously for 30 minutes, five times a week.
  Arms: Bilateral iTNS; Unilateral iTNS
Device: Sham iTNS — The sham devices are designed to mimic active stimulation by initially delivering electrical current sufficient to evoke toe flexion. However, once the current is reduced to the sensory stimulation threshold, the device automatically ramps down to 0mA while maintaining the appearance of normal functioning on the display screen.
  Arms: Sham iTNS; Unilateral iTNS

SUMMARY:
The purpose of this study is to determine the safety and efficacy of Injectrode Tibial Nerve Stimulation for bladder function in people with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Non-progressive chronic (>1 year) SCI
* Neurologic level of injury T9 and above
* Stable over active bladder (OAB) medications (≥3 months)
* No contraindication to MRI (per MRI Safety Questionnaire)
* English or Spanish speaking
* Tolerate and be able to evoke toe flexion bilaterally with transcutaneous tibial nerve stimulation (tTNS) (self or assisted)
* Pass the tTNS competency checklist to perform or direct performance of tTNS.

Exclusion Criteria:

* Ongoing/active genitourinary oncologic diagnoses
* History of other central nervous system disorder (CNS) disorders and/or peripheral neuropathy
* Pregnancy or planning to become pregnant.
* Lower Motor Neuron bladder
* Restorative bladder surgery such as augmentation cystoplasty
* Botulinum toxin-A injections in the bladder within 6 months of trial enrolment (injection in other sites is allowed)
* Anticoagulation treatment or prophylaxis
* Advanced peripheral vascular disease (gangrene, amputation, etc.)
* History of intolerance to electrical stimulation, particularly of the leg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by the number of device-related adverse events | From baseline to 8 weeks
  Adverse events include lead migration and fracture, hematoma, wound infection, delayed healing, nerve injury, and autonomic dysreflexia occurrence during the procedure.
Accuracy as assessed by the percentage of sessions where toe flexion was achieved as recorded in subject logs. | From baseline to week 8
Reliability as assessed by the average minimum current (mA) required to elicit toe flexion when testing for accuracy | From baseline to week 8
Feasibility of Injectrode procedure as assessed by surveys | Week 8
  Feasibility to check if reproducible training pathway can enable non-interventional physicians to competently perform Injectrode implantation and removal
Physician acceptability of Injectrode device as assessed by a survey | Week 8
  The acceptability survey ranges from 0 - 32, with a higher score indicating greater acceptability of the Injectrode device.
Participant acceptability of Injectrode device as assessed by a survey | Week 8
  The acceptability survey ranges from 0 - 25, with a higher score indicating greater acceptability of the Injectrode device.
Feasibility and acceptability of the Injectrode treatment as assessed by a qualitative interview | Week 8
  A semi-structured interview will be conducted with participants and providers to explore their perceptions of the Injectrode treatment. Responses will be summarized using qualitative coding and descriptive statistics of themes.

SECONDARY OUTCOMES:
Number of participants for whom bladder medication dosage reduced | from baseline to 8 weeks
Change in magnitude of dosage of medication | from baseline to 8 weeks
Change in bladder function during urodynamics as assessed by the maximum detrusor pressure (Max Pdet) in cmH20. | Baseline, Week 4, and Week 8
Change in Bladder function as assessed by the presence or absence of detrusor overactivity (DO) during urodynamics. | baseline, Week 4, and Week 8
Change in bladder capacity (maximum volume in mL) during urodynamics before voiding or discomfort. | baseline, Week 4, and Week 8
Change in the presence or absence of leaks during urodynamics. | baseline, Week 4, and Week 8
Change in bladder sensation during urodynamics as defined by the infused volume (mL) at time of reported first sensation of filling. | baseline, Week 4, and Week 8
Change in bladder sensation during urodynamics as defined by infused volume (mL) at time of reported urgency/ desire to void. | Baseline, Week 4, and Week 8
Change in bladder sensation during urodynamics as defined by the infused volume (mL) at the time of reported discomfort. | Baseline, Week 4, and Week 8
Change in detrusor compliance during urodynamics as reported by the change in bladder volume divided by the change in bladder pressure. | baseline, Week 4, and Week 8
Change in the number of incontinence episodes as self-reported in the bladder diary. | Baseline, Week 4, and Week 8
Change in the frequency of catheterization as self-reported in the bladder diary. | Baseline, Week 4, and Week 8
Change in the volume of catheterization as self-reported in the bladder diary. | Baseline, Week 4, and Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Argyrios Stampas, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No